CLINICAL TRIAL: NCT04805736
Title: A Pilot Study of Single-Dose Camrelizumab and/or Microwave Ablation in Women With Early-Stage Breast Cancer
Brief Title: Microwave Ablation Combined With Camrelizumab in the Treatment of Early Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shui Wang, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-Ⅱ-021
Record Dates: First submitted 2021-03-10; First posted 2021-03-18 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: Ablation; PD-1; Immunotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — camrelizumab; Mastectomy, Segmental

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Microwave Ablation alone (Experimental): Microwave Ablation+ Breast Surgery
  Interventions: Procedure: Microwave Ablation; Procedure: Breast Surgery
- Camrelizumab alone (Experimental): Camrelizumab+ Breast Surgery
  Interventions: Drug: Camrelizumab; Procedure: Breast Surgery
- Microwave Ablation & Camrelizumab (Experimental): Microwave Ablation + Camrelizumab + Breast Surgery
  Interventions: Procedure: Microwave Ablation; Drug: Camrelizumab; Procedure: Breast Surgery

INTERVENTIONS:
Procedure: Microwave Ablation — Image-guided microwave ablation 7-10 days prior to surgery
  Arms: Microwave Ablation & Camrelizumab; Microwave Ablation alone
Drug: Camrelizumab — Camrelizumab 200 mg was given a few days after microwave ablation
  Other Names: SHR-1210
  Arms: Camrelizumab alone; Microwave Ablation & Camrelizumab
Procedure: Breast Surgery — Standard of care breast conserving surgery or radical mastectmoy

SUMMARY:
Ablative therapy, as a local treatment modality for tumors, has an immune activating effect. To explore the synergistic effect of microwave ablation combined with PD-1 inhibitors, this prospective, open-label, multi-cohort, single-center clinical study was conducted. To compare the feasibility and safety of preoperative microwave ablation alone, with or without camrelizumab in patients with early newly diagnosed breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female.
2. Age 20-65 years.
3. Invasive carcinoma confirmed by core biopsy.
4. Newly diagnosed breast cancer patients, without adjuvant therapy.
5. Imaging findings showed a single breast tumor with a maximum diameter of 3 cm, no distant metastasis, and no invasion of the skin and chest wall.
6. Systematic ultrasound is able to visualize lesions.
7. Surgical treatment was planned.
8. The functional level of major organs must meet the following requirements:

   1. blood routine: neutrophil (ANC) ≥ 1.5 × 109/L; platelet count (PLT) ≥ 90 × 109/L; hemoglobin (Hb) ≥ 90 g/L;
   2. blood biochemistry: total bilirubin (TBIL) ≤ upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × ULN; alkaline phosphatase ≤ 2.5 × ULN; blood urea nitrogen (BUN) and creatinine (Cr) ≤ 1.5 × ULN;
   3. coagulation: international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN; activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
   4. Heart: left ventricular ejection fraction (LVEF) ≥ 50% as assessed by echocardiography (ECHO) or multigated acquisition (MUGA).
   5. Thyroid function: thyroid stimulating hormone (TSH) ≤ ULN; if abnormal, T3 and T4 levels should be investigated, and normal T3 and T4 levels can be included.
   6. Urinalysis: urine protein < 2 +, if urine protein ≥ 2 +, 24-hour urine protein quantification must show protein ≤ 1 g.
9. Voluntarily participate in this study, sign informed consent, have good compliance and are willing to cooperate with follow-up.

Exclusion Criteria:

1. Tumor involving skin, ulceration, inflammatory breast cancer patients
2. Fatty breast cancer.
3. Tumors on the deep surface of areolar region
4. KPS score < 70, or ECOG score > 2
5. Patients with a history of concomitant collagen connective tissue disease, or any active autoimmune disease or autoimmune disease.
6. Prior radiotherapy or prior use of investigational drugs or other immunosuppressive agents
7. Heart, brain, lung, kidney and other vital organ failure, liver and kidney dysfunction;
8. Uncorrectable severe coagulopathy
9. Patient is pregnant or lactating
10. Poor glycemic control in diabetes
11. Patients with foreign body implantation around the tumor
12. Patients with severe scars on the skin of the treatment area (protruding from the skin surface, width ≥ 1 cm)
13. History of chronic immunosuppression, prior immunotherapy, recent vaccination (< 4 weeks)
14. Human immunodeficiency virus (HIV) infection, active hepatitis B (hepatitis B indicates antigen positive and HBV DNA ≥ 500 IU/ml), hepatitis C (hepatitis C antibody positive and HCV-RNA above the lower limit of detection of the analytical method).
15. Concurrent medical conditions that, in the judgment of the investigator, would jeopardize the subject's safety, could confound the study results, or affect the subject's completion of this study.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Safety of Microwave Ablation Combined With Camrelizumab | 3 months
  Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 5.0

SECONDARY OUTCOMES:
Complete ablation rate | 1 day
  The proportion of patients with complete ablation was calculated for all patients. Complete ablation was defined as: tissue section at the ablation margin that was negative by histochemical staining.
Negative predictive value of ultrasound | 1 day
  Preoperative ultrasonography was performed. The negative predictive value of ultrasound was calculated by comparing the pathology report. Negative predictive value = number of patients with negative pathology and negative ultrasound/number of patients with negative ultrasound
Assessment of Immunogenicity | 3 months
  Proportion of subjects with immune response to synergistic therapy detected by biomarkers in peripheral blood samples
Breast self evaluation | 3 months
  Breast self evaluation for patients will be assessed by Functional Assessment of Cancer Therapy - Breast (FACT-B) scale scores.The FACT-B consists of 44 self-report items and assesses the specific breast cancer-related quality of life on 4 general and 1 breast-cancer specific subscale. A higher score indicates a higher cancer-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Available from the corresponding author upon reasonable request
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Pan H, Yu M, Tang X, Mao X, Liu M, Zhang K, Qian C, Wang J, Xie H, Qiu W, Ding Q, Wang S, Zhou W. Preoperative single-dose camrelizumab and/or microwave ablation in women with early-stage breast cancer: A window-of-opportunity trial. Med. 2024 Apr 12;5(4):291-310.e5. doi: 10.1016/j.medj.2024.01.015. Epub 2024 Feb 27. PMID 38417440